CLINICAL TRIAL: NCT05605730
Title: Maitland Thoracic Mobilization Versus Mulligan Thoracic Mobilization in Kyphotic Patients With Shoulder Impingement Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mahmoud Salah Yousef Aboraya, Assistant lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/003447
Record Dates: First submitted 2022-10-30; First posted 2022-11-04 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2024-01

CONDITIONS: Shoulder Impingement Syndrome; Kyphosis Thoracic
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Traditional exercise management (Active Comparator): 1. Prone back extension.
  2. Shoulder external rotation starting in 45° of internal rotation, with the arm by the side and the elbow flexed to 90 °.
  3. Shoulder internal rotation starting in 45 ° of external rotation, with the arm by the side and the elbow flexed to 90 °..
  4. Shoulder abduction (scapular plane) through a 0- to 60-° with the elbow flexed 90 ° and the shoulder in neutral rotation.
  5. Shoulder flexion (sagittal plane) through a 0- to 60-°starting with the elbow flexed 90 ° and the shoulder in neutral rotation and punching forward, simultaneously extending the elbow and flexing the shoulder.
  6. Internal rotation towel stretch: Subjects will be instructed to sit or stand while holding a towel with the affected arm behind the back and to use the other arm to pull the affected arm up the back.
  Interventions: Other: Traditional exercise management
- Maitland mobilization for thoracic spine (Experimental): This group will receive the previously mentioned exercises protocol targeting shoulder joint in addition to Maitland mobilization for thoracic spine.
  Interventions: Other: Maitland mobilization for thoracic spine; Other: Traditional exercise management
- Mulligan thoracic sustained natural apophyseal glide (SNAGS) (Experimental): Treatment would be administered at the vertebral level revealed during the evaluation of thoracic SNAG.
  Interventions: Other: Mulligan thoracic sustained natural apophyseal glide (SNAGS); Other: Traditional exercise management

INTERVENTIONS:
Other: Maitland mobilization for thoracic spine — The thoracic spine mobilization will be consisting of oscillations to the thoracic vertebrae from the prone positions for repeated 30 times with 1 min interval between each 4 sets for 15 minutes. For central posterio-anterior mobilization, a grade III large amplitude rhythmic oscillation in the postero-anterior direction will be applied to the joint sign segment which is defined as the patient's most painful or hardest to move segment. It will be detected through a passive accessory intervertebral motion (PAIVM) test. T6,7 will be used as a site for application if the joint sign can't be detected. The frequency of treatment sessions will be 3 sessions per week for 4 weeks.
  Arms: Maitland mobilization for thoracic spine
Other: Mulligan thoracic sustained natural apophyseal glide (SNAGS) — Verbal instructions will be provided for the patient to move into thoracic extension and do over-pressure at the end of ROM while a transverse glide is maintained by the therapist for a set of 10 repetitions. The significance of performing a pain-free movement will be emphasized to the patient all the time. There will be 3 sets of 10 repetitions with one minute rest between each set.
  Arms: Mulligan thoracic sustained natural apophyseal glide (SNAGS)
Other: Traditional exercise management — Prone back extension. Shoulder external rotation starting in 45° of internal rotation, with the arm by the side and the elbow flexed to 90 °.
  Shoulder internal rotation starting in 45 ° of external rotation, with the arm by the side and the elbow flexed to 90 °..
  Shoulder abduction (scapular plane) through a 0- to 60-° with the elbow flexed 90 ° and the shoulder in neutral rotation.
  Shoulder flexion (sagittal plane) through a 0- to 60-°starting with the elbow flexed 90 ° and the shoulder in neutral rotation and punching forward, simultaneously extending the elbow and flexing the shoulder.
  Internal rotation towel stretch: Subjects will be instructed to sit or stand while holding a towel with the affected arm behind the back and to use the other arm to pull the affected arm up the back.

SUMMARY:
In recent years the management of shoulder impingement syndrome (SIS) included the thoracic spine as it was proved that it's highly correlated to pathologies in shoulder joint. SIS is proved to be associated with kyphotic posture. Also, It was proved that changing sitting posture affects the measured ROM of shoulder joint and this implicates the influence of changing thoracic position on shoulder mechanics. Explanations were made regarding the role of thoracic spine in affecting the shoulder joint through two ways. Firstly, through affecting the mechanics of scapular movements and secondly through altering the length tension relationship of shoulder musculature. This study would aim at studying the most effective thoracic mobilization in the treatment of SIS.

ELIGIBILITY:
Inclusion Criteria:

* Shoulder impingement syndrome SIS clinically diagnosed by using Hawkins-Kennedy test, the painful arc test, and the infraspinatus muscle strength test; and for a rotator cuff tear, the infraspinatus and the drop-arm test and supraspinatus muscle strength tests.
* Subjects will be diagnosed of having postural kyphosis proved by a physician referral or modified Cobb's angle of more than 40 degrees (x-ray).

Exclusion Criteria:

* The participants with any musculoskeletal abnormalities eg. Glenohumeral instability.
* Neurological abnormalities.
* Surgical operation of the last 4 months will be excluded from the study.
* Shoulder corticosteroid injection at any time in the past.
* Engaging in any athletic physical activities.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-04 (Actual); Primary Completion 2023-09-14 (Actual); Study Completion 2023-12-20 (Actual)

PRIMARY OUTCOMES:
Active ROM of shoulder joint would be measured utilizing goniometric method | 6 weeks
  The patient will move the affected shoulder with the thumb pointing upwards through the full available active range of shoulder flexion, abduction and external rotation. The flexion angle will be formed by aligning the goniometer with the lateral epicondyle of the humerus, a vertical line in the coronal plane and the axis with the middle of the glenoid fossa. The abduction angle will be formed by aligning the goniometer with the lateral epicondyle of the humerus, a vertical line in the sagittal plane , and the axis in the middle of the posterior glenohumeral joint line. The external rotation angle will be formed by aligning the goniometer with the ulna styloid process, a horizontal line in the transverse plane , and the axis at the olecranon process of the ulna.
Kyphotic angle utilizing photographic method | 6 weeks
  A lateral view image of the patient will be analyzed after fitting lateral earlobe markers. The patient will stand sideways against a calibration plane with shoulders and elbows at flexed 90 degrees while looking at a fixed point on the opposite wall. The shooting will be repeated 3 times with a camera placed 1.5 meters away from the calibration plane and at a one-meter height from the ground on a tripod. In the software, a line parallel to the calibration plane from the ear lobe would be considered the plumb line. The farthest point from the plumb line will be considered the apex of the kyphosis angle. Then, two lines at the top and bottom running parallel to the curvature of the back are considered the two lines of the angle. These lines intersected at the apex of each other. The angle of intersection of the lines was measured by Kinovea and decreased from 180°.
The Arabic version of the Disability of Arm, Shoulder and Hand (DASH-Arabic) | 6 weeks
  The DASH-Arabic contains 30 items relating to the level of difficulty the patient faces while performing different activities using the arm, shoulder and hand; items assessing the severity of pain symptoms; and items assessing problems that affect social activities, work and sleep, and psychological impact. In the DASH-Arabic, each item has five response choices that range from 1, ''without any difficulty or no symptoms exist'' to 5, ''unable to engage in activity or very severe symptoms''. A minimum of 27 of the 30 items must be completed for the questionnaire to be regarded. The higher the score, the greater the disability.
Pain will be assessed using visual analogue scale. | 6 weeks
  Scores are based on self-reported measures of symptoms that are recorded with a single handwritten mark placed at one point along the length of a 10-cm line that represents a continuum between the two ends of the scale-"no pain" on the left end (0 cm) of the scale and the "worst pain" on the right end of the scale (10 cm)

CONTACTS AND LOCATIONS:
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No